CLINICAL TRIAL: NCT06107426
Title: A Global Real-World Evidence Study on the Long-term Effectiveness of ABBV-951 in Advanced Parkinson´s Disease in Routine Clinical Practice (ROSSINI: Real-world Outcomes With continuouS Subcutaneous Levodopa INfusIon)
Brief Title: Real-World Study of ABBV-951 Subcutaneous Infusion to Assess Change in Disease Activity in Adult Participants With Parkinson's Disease
Acronym: ROSSINI
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-487
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease; Advance Parkinson's Disease; ABBV-951; Foslevodopa/foscarbidopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A: ABBV-951: Participants naïve to ABBV-951 will receive ABBV-951 as prescribed by their physician according to the local label.
- Cohort B: ABBV-951: Participants transitioning from the Open-Label Extension studies M15-737 and M20-098 will continue to receive ABBV-951.
- Country Specific Sub-Study: Participants located in the United States, Germany and Spain, that participated in Cohort A, will participate in a single initial interview and those who continue on the treatment after 6 months will participate in a follow-up interview to explore the longitudinal impact of the treatment. Those participants who discontinue prior to the 6 months time point will engage in a discontinuation interview to understand reasons for their discontinuation of treatment.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. The purpose of this study is to evaluate how effective ABBV-951 is in treating adult participants with advanced PD in real world setting.

ABBV-951 (foslevodopa/foscarbidopa) is an approved drug for the treatment of Parkinson's Disease. The main ROSSINI study will have approximately 450 adult participants with PD (300 participants new to ABBV-951, up to 150 participants transitioning from open-label extension study) will be enrolled across approximately 60 sites. Decision to treat with ABBV-951 (or continue the treatment in Cohort B) will be made by the doctor prior to any decision to approach the participant to participate in this study. There will be a sub-study that will enroll 40 naïve participants who initiated Foslevodopa/Foscarbidopa treatment for the first time (Cohort A of the ROSSINI parent study only) from 6 to 15 centers in the United States, Germany and Spain.

All participants will receive subcutaneous infusion of ABBV-951 for approximately 3 years.

Participants will attend regular clinic visits during the course of the study. The effect of the treatment will be checked by medical assessments, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for ABBV-951 therapy in accordance with the approved local label in the participating country and local reimbursement regulations, if applicable.
* Diagnosis of levodopa-responsive idiopathic Parkinson's Disease (PD).
* Participant must be either:

  * Cohort A: Naïve to ABBV-951
  * Cohort B: Pre-treated with ABBV-951, specifically, participants of Open-Label Extension Studies M15-737 and M20-098 who completed these studies without significant protocol deviations and who did not experience an adverse event (AE) that in the investigator's opinion may indicate an unacceptable safety risk.
* Decision to treat with ABBV-951 (or continue the treatment in Cohort B) made by the clinician prior to any decision to approach the participant to participate in this study.
* Prior to any study-related procedures being performed, the participant, or legal authorized representative (LAR) has voluntarily signed an Authorization for Use/Disclosure of Data (AUDD)/informed consent form (ICF) according to national regulations after the study has been explained and the participant has had the opportunity to have questions answered.

Exclusion Criteria:

* Any condition included in the contraindications section of the approved local ABBV-951 label in the participating country.
* Mini-Mental State Examination (MMSE) score < 24.

  * If the participant has a score of 19-23, he/she can be included if based on the investigator´s judgment the participant is able to handle the therapy and follow the study procedures with the help of a permanent caregiver.
* Participation in a concurrent interventional clinical trial from enrollment and throughout the study.
* History of significant skin conditions or disorders per investigator´s judgment. In case of temporary affections like recent sunburn, acne, scar tissue, tattoo, open wound, branding, or colorations, the participant should not be included if the investigator considers these as interfering with the infusion of study drug or with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Advanced PD, treated with ABBV-951 according to label and local reimbursement regulations, where applicable.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in OFF Time (hours) | Up to approximately 3 years
  The mean change from baseline to each scheduled visit in the number of hours spent in OFF time will be estimated using a mixed-effect model repeated-measures (MMRM).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (68):
- United States (27):
  - University of Alabama at Birmingham - Main /ID# 253477, Birmingham, Alabama
  - Banner Sun Health Research Institute /ID# 253461, Sun City, Arizona
  - Parkinson's Research Centers of America - Palo Alto /ID# 264703, Palo Alto, California
  - Georgetown University Hospital /ID# 259381, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton /ID# 253465, Boca Raton, Florida
  - University of Florida College of Medicine /ID# 259383, Gainesville, Florida
  - University of Miami /ID# 259396, Miami, Florida
  - N1 Research, LLC /ID# 264221, Orlando, Florida
  - University of South Florida- Neuroscience Institute /ID# 253470, Tampa, Florida
  - Northwestern Medicine Primary And Specialty Care Lavin Family Pavilion /ID# 266977, Chicago, Illinois
  - Ochsner Medical Center - Jefferson Highway /ID# 269764, New Orleans, Louisiana
  - Boston Medical Center Health System /ID# 269765, Brighton, Massachusetts
  - University of Minnesota - Minneapolis /ID# 268121, Minneapolis, Minnesota
  - Kansas City VA Medical Center /ID# 253466, Kansas City, Missouri
  - Cleveland Clinic Lou Ruvo Cent /ID# 259390, Las Vegas, Nevada
  - David L. Kreitzman, MD, PC /ID# 259397, Commack, New York
  - Northwell Health /ID# 253469, Lake Success, New York
  - Novant Health Neurology and Sleep /ID# 259391, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 259387, Winston-Salem, North Carolina
  - NeuroCare Center /ID# 259392, Canton, Ohio
  - The Movement Disorder Clinic of Oklahoma /ID# 253463, Tulsa, Oklahoma
  - Vanderbilt University Medical Center /ID# 253474, Nashville, Tennessee
  - Texas Movement Disorder Specialists /ID# 253473, Georgetown, Texas
  - Univ Texas HSC San Antonio /ID# 259394, San Antonio, Texas
  - University of Utah /ID# 253471, Salt Lake City, Utah
  - Evergreenhealth Medical Center /ID# 268120, Kirkland, Washington
  - Inland Northwest Research /ID# 253460, Spokane, Washington
- Australia (2):
  - Westmead Hospital /ID# 259670, Westmead, New South Wales
  - The Royal Melbourne Hospital /ID# 259671, Parkville, Victoria
- Austria (4):
  - Medizinische Universitaet Graz /ID# 262774, Graz, Styria
  - Medizinische Universitaet Innsbruck /ID# 262775, Innsbruck, Tyrol
  - Kepler Universitaetsklinikum GmbH /ID# 262776, Linz, Upper Austria
  - Klinik Ottakring /ID# 262773, Vienna, Vienna
- Canada (4):
  - University of Calgary /ID# 262833, Calgary, Alberta
  - The Ottawa Hospital - General Campus /ID# 263315, Ottawa, Ontario
  - CHUM - Centre hospitalier de l'Universite de Montréal /ID# 269689, Montreal, Quebec
  - Centre de Recherche St-Louis /ID# 262746, Québec, Quebec
- Denmark (3):
  - Bispebjerg Hospital /ID# 252032, Copenhagen, Capital Region
  - Rigshospitalet Glostrup /ID# 252035, Glostrup Municipality, Capital Region
  - Odense University Hospital /ID# 252036, Odense, Region Syddanmark
- Germany (7):
  - Parkinson-Klinik Ortenau GmbH&Co KG /ID# 252376, Wolfach, Baden-Wurttemberg
  - Klinikum der Universitaet Muenchen Grosshadern /ID# 255574, Munich, Bavaria
  - Klinikum Ernst von Bergmann /ID# 252375, Potsdam, Brandenburg
  - Klinikum Osnabrueck GmbH /ID# 252275, Osnabrück, Lower Saxony
  - Krankenhaus Martha-Maria Halle-Doelau /ID# 260372, Halle, Saxony-Anhalt
  - Kliniken Beelitz GmbH /ID# 252665, Beelitz-Heilstätten
  - Knappschaftskrankenhaus Bottrop /ID# 252274, Bottrop
- Israel (6):
  - Shaare Zedek Medical Center /ID# 257715, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 254823, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 254824, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 260421, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 257717, Jerusalem
  - Rabin Medical Center. /ID# 257716, Petah Tikva
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Timisoara /Id# 252248, Timișoara, Timiș County
  - Spitalul Clinic Judetean de Urgenta Timisoara /Id# 252249, Timișoara, Timiș County
  - Spitalul Clinic Judetean de Urgenta Brasov /ID# 253308, Brasov
  - Spitalul Clinic Colentina /ID# 252250, Bucharest
  - Spitalul Clinic Judetean de Urgenta Constanta /ID# 252251, Constanța
  - Spitalul Clinic Judetean de Urgenta Targu Mures /ID# 252247, Târgu Mureş
- Spain (6):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 261402, Santiago de Compostela, A Coruna
  - Hospital General Universitario de Elche /ID# 254438, Elche, Alicante
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 260921, Majadahonda, Madrid
  - Hospital Universitario Virgen de las Nieves /ID# 257588, Granada
  - Hospital Clinico San Carlos /ID# 260922, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 254437, Seville
- Sweden (3):
  - Centrum for neurologi /ID# 252118, Stockholm, Stockholm County
  - Uppsala University Hospital /ID# 252119, Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset /ID# 252115, Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P22-487